CLINICAL TRIAL: NCT04398628
Title: ATHN Transcends: A Natural History Cohort Study of the Safety, Effectiveness, and Practice of Treatment in People With Non-Neoplastic Hematologic Disorders
Brief Title: ATHN Transcends: A Natural History Study of Non-Neoplastic Hematologic Disorders
Status: Recruiting | Type: Observational
Sponsor: American Thrombosis and Hemostasis Network (Network)
Collaborators: Pfizer (Industry); Hemophilia of Georgia, Inc. (Other); Genentech, Inc. (Industry); CSL Behring (Industry); Sanofi (Industry); Novo Nordisk A/S (Industry); Hemab ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: ATHN Transcends
Record Dates: First submitted 2020-05-11; First posted 2020-05-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Disorder; Bleeding Disorder; Connective Tissue Disorder; Hemophilia; Thrombosis; Von Willebrand Diseases; Thrombophilia; Rare Bleeding Disorder; Platelet Disorder; Factor IX Deficiency; Factor VIII Deficiency; Thalassemia; Sickle Cell Disease
MeSH Terms: conditions — Hematologic Diseases; Hemostatic Disorders; Connective Tissue Diseases; Hemophilia A; Thrombosis; von Willebrand Diseases; Thrombophilia; Blood Platelet Disorders; Hemophilia B; Thalassemia; Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All participants have the option to provide consent to have specimens stored in the ATHN Transcends Biorepository.
  Inhibitor titer testing will be performed locally (unless otherwise specified) as per standard of care which is generally expected to coincide with the following:
  * Baseline Visit
  * Annual Visit
  * Product switch
  * Suspected inhibitor development
  * Confirmatory test for previously elevated result
  * Study Exit
  * Additional timepoints per any modules
  Genetic testing (performed once) will be optional and provided by central labs, as funding allows, across all cohorts.
  Anti-drug antibodies testing - For participants receiving non-factor products (e.g., emicizumab) and if testing is clinically appropriate (suspicion of anti-drug antibodies forming), this specimen will be analyzed, as funding allows.
  Factor activity testing will be performed locally at the following timepoints:
  * Baseline visit
  * 6 and 18-month follow-up visits
  * Annual visit
  * Ad hoc
  * Study arm exit
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Hemophilia: This cohort includes three Arms and six Modules:
  Previously Untreated Patients (PUPs) Arm
  Efanestoctocog alfa (ALTUVIIIO®) Module
  INHIBIT Module
  Hemophilia Natural History Arm
  Emicizumab (Hemlibra®) Module
  Nonacog beta pegol (Rebinyn®)Module
  Distress Module
  Hemophilia Gene Therapy Outcomes Arm
  Etranacogene dezaparvovec (HEMGENIX®) Module
- Congenital Platelet Disorders: This cohort includes one Arm and Module:
  Congenital Platelet Disorders (CPD) Natural History Arm Glanzmann Thrombasthenia (GT) Module
- Von Willebrand Disease: No arms or modules
- Rare Disorders: No arms or modules
- Bleeding NOS: No arms or modules
- Thrombosis/Thrombophilia: No arms or modules
- Non-Neoplastic Hematologic Conditions: No arms or modules

SUMMARY:
In parallel with the growth of ATHN's clinical studies, the number of new therapies for all blood disorders is increasing significantly. Some of the recently FDA-approved therapies for congenital and acquired hematologic conditions have not yet demonstrated long-term safety and effectiveness beyond the pivotal trials that led to their approval. In addition, results from well controlled, pivotal studies often cannot be replicated once a therapy has been approved for general use.2,3,4,5

In 2019 alone, the FDA has issued approvals for 24 new therapies for congenital and acquired hematologic conditions.6 In addition, almost 10,000 new studies for hematologic diseases are currently registered on www.clinicaltrials.gov.7

With this increase in potential new therapies possible, it is imperative that clinicians and clinical researchers in the field of non-neoplastic hematology have a uniform, secure, unbiased, and enduring method to collect long-term safety and efficacy data. As emphasized in a recently published review, accurate, uniform and quality national data collection is critical in clinical research, particularly for longitudinal cohort studies covering a lifetime of biologic risk.8

DETAILED DESCRIPTION:
This is a longitudinal, natural history observational cohort study being conducted at approximately 150 ATHN-affiliated sites with a target accrual of 3,000 participants. Participants will be followed for a minimum of 15 years on an assigned arm within a cohort; however, arm or module participation may last longer, and participants will continue participation in the arm or module for its duration. Harmonized data elements will be collected at the time of enrollment, semi-annually (every 6 months), annually, ad hoc, and as defined by the terms of individual arms and modules. Data will be collected for participants enrolled in cohort-specific arms and modules.

Each participant will be assigned to a single cohort: Hemophilia, von Willebrand Disease, Congenital Platelet Disorders, Rare Disorders, Bleeding Not Otherwise Specified (NOS), Thrombosis/Thrombophilia, or Non-Neoplastic Hematologic Conditions.

Study arms and study modules are developed to advance the exploration of blood disorders disease specific insights by ATHN and its partners. Arms may branch off into product-specific data collection via Modules to be collected during the study, in conjunction with planned study assessments.

ATHN Transcends

Co- Principal Investigators:

Tammuella Chrisentery-Singleton, MD Ochsner Clinic Foundation American Thrombosis and Hemostasis Network

Michael Recht, MD, PhD, MBA Yale University School of Medicine National Bleeding Disorders Foundation

PUPs Arm

Principal Investigator:

Shannon Carpenter, MD, MS University of Missouri Kansas City School of Medicine Children's Mercy Hospital

ALTUVIIO Module

Principal Investigator:

Shannon Carpenter, MD, MS University of Missouri Kansas City School of Medicine Children's Mercy Hospital

INHIBIT Module

Principal Investigator:

Nicoletta Machin DO, MS Hemophilia Center of Western Pennsylvania University of Pittsburgh Medical Center

Hemophilia Natural History Arm

Principal Investigator:

Fernando Corrales-Medina, MD, FAAP University of Miami-Comprehensive Hemophilia Treatment Center University of Miami-Miller School of Medicine

Rebinyn Module

Co-Principal Investigators:

Lauren Amos, MD University of Missouri Kansas City School of Medicine Children's Mercy Hospital

Guy Young, MD University of Southern California Children's Hospital Los Angeles

Distress Module

Principal Investigator:

Tammuella Chrisentery-Singleton, MD Ochsner Clinic Foundation American Thrombosis and Hemostasis Network

Hemlibra Module

Principal Investigator:

Fernando Corrales-Medina, MD, FAAP University of Miami-Comprehensive Hemophilia Treatment Center University of Miami-Miller School of Medicine

Hemophilia Gene Therapy Outcomes Arm:

Co-Principal Investigators:

Janice M. Staber, MD Iowa Hemophilia and Thrombosis Center University of Iowa Stead Family Children's Hospital

Ulrike M. Reiss, MD Hemophilia Treatment Center St. Jude's Children's Research Hospital

HEMGENIX Module

Co-Principal Investigators:

Janice M. Staber, MD Iowa Hemophilia and Thrombosis Center University of Iowa Stead Family Children's Hospital

Ulrike M. Reiss, MD Hemophilia Treatment Center, St. Jude's Children's Research Hospital

Severe VWD Natural History Arm:

Co-Principal Investigators:

Robert F. Sidonio, Jr., MD, MSc Aflac Cancer and Blood Disorders Center, Hemophilia of Georgia Center for Bleeding and Clotting Disorders

Angela C. Weyand, MD C.S. Mott Children's Hospital, University of Michigan Medical School, Ann Arbor

Congenital Platelet Disorders Natural History Arm:

Principal Investigator Sanjay Ahuja, MD Innovative Hematology, Indiana Hemophilia & Thrombosis Center

Glanzmann Thrombasthenia Module:

Co-Principal Investigators:

Divya Citla-Sridhar, MD University of Arkansas for Medical Sciences Arkansas Children's Hospital

Meera Chitlur, MD Central Michigan University, Children's Hospital of Michigan

Hemophilia Cohort

This cohort includes three Arms and six Modules:

Previously Untreated Patients (PUPs) Arm This is a pediatric focused Arm of PUPs with hemophilia A or B of any severity.

Efanestoctocog alfa (ALTUVIIIO®) Module The purpose is to investigate the safety, tolerability, and effectiveness of efanesoctocog alfa (ALTUVIIIO®) in PUPs with severe hemophilia A.

INHIBIT Module This is an observational study assessing the rate of inhibitor formation in young children with severe hemophilia A in the current treatment era.

Hemophilia Natural History Arm This Arm is investigating the safety, effectiveness, and practice of treatment for people with hemophilia.

Emicizumab (Hemlibra®) Module All participants treated with Hemlibra® are eligible to participate.

Distress Module Participants with Congenital Hemophilia A or B, 18 years of age or older, will be followed longitudinally for 2 years or from time of enrollment for a total planned study duration of 3 years

Nonacog beta pegol (Rebinyn®) Module The Rebinyn® Module is a prospective study in hemophilia B participants without inhibitors.

Hemophilia Gene Therapy Outcomes Arm This Arm is investigating the safety and effectiveness of gene therapy in people with hemophilia.

Etranacogene dezaparvovec (HEMGENIX®) Module This is an observational study to characterize the effectiveness and safety of HEMGENIX® in participants with hemophilia B.

Congenital Platelet Disorders (CPD) Natural History Arm:

The CPD Arm is investigating the natural history of the safety and efficacy of hemostatic therapies (such as platelet transfusions, desmopressin, antifibrinolytics, recombinant factor VIIa) in the prevention or treatment of bleeding events (on demand, surgery, prophylaxis) in adult and pediatric participants with inherited congenital platelet disorders..

Glanzmann Thrombasthenia (GT) Module:

This Module is a study of bleeding symptoms, treatments, and treatment outcomes in patients with Glanzmann thrombasthenia.

Von Willebrand Disease Cohort No arms or modules open at this time.

Rare Disorders Cohort No arms or modules open at this time.

Bleeding NOS No arms or modules open at this time.

Thrombosis/Thrombophilia No arms or modules open at this time.

Non-Neoplastic Hematologic Conditions No arms or modules open at this time.

ELIGIBILITY:
Participants who meet the following inclusion criteria and none of the exclusion criteria are eligible for enrollment in one of the open disease-specific arms.

Inclusion Criteria:

1. Any age
2. Having a congenital or acquired blood disorder; or
3. Having a bleeding phenotype as indicated by an age adjusted abnormal ISTH Bleeding Assessment Tool score with an unknown diagnosis; or
4. Connective tissue disorder with bleeding tendency as indicated by an age adjusted abnormal ISTH Bleeding Assessment Tool score.
5. Eligible for a currently active disease-specific arm.
6. Concurrent enrollment in the ATHNdataset or current ATHNdataset participant.

Exclusion Criteria:

1. Does not qualify for inclusion in a currently activedisease-specific arm; participants may be eligible to enroll as future cohorts and arms are activated; 2. Unable to give informed consent or assent 3. Unwilling to perform study procedures

Cohort Participant Selection

Each participant is to be enrolled in the cohort for which they qualify as defined below.

Hemophilia Cohort

Inclusion Criteria:

Participants who meet any of the following inclusion criteria are eligible for enrollment into this cohort:

1. Factor VIII or factor IX activity <50%, without another explanation for low clotting factor other than congenital hemophilia or being a known carrier for congenital hemophilia; OR
2. Carrier for congenital hemophilia with a factor VIII >=50% or factor IX activity >=50% with or without a bleeding phenotype as indicated by an ISTH Bleeding Assessment Tool score of ≥4 for adult males, ≥6 for adult females, or ≥3 for children younger than 18 years OR
3. Known congenital hemophilia that have a factor level >50% after receiving vector, OR 4. Acquired hemophilia.

Exclusion Criteria:

None

Von Willebrand Disease Cohort

Inclusion Criteria:

Participants who meet the following inclusion criteria are eligible for enrollment into this cohort:

1. Meeting the definition of VWD or low VWF per most recent international guidelines

Exclusion Criteria:

None

Congenital Platelet Disorders Cohort

Inclusion Criteria:

Participants who meet the following inclusion criteria are eligible for enrollment into this cohort:

1. Abnormalities of platelet function a. Glanzmann thrombasthenia (GPIIb or GPIIIa) b. Bernard-Soulier syndrome (GPIbalpha, GPIbbeta, or GPIX)
2. Abnormalities of platelet granules
3. Abnormalities of platelet signal transduction
4. Abnormalities of platelet secretion
5. Collagen Receptor Defect
6. ADP Receptor Defect
7. Thromboxane Receptor Defect
8. Giant Platelet Disorder
9. Abnormalities in platelet aggregation testing due to another or unknown cause (not drug related)

Exclusion Criteria:

1. Platelet disorders secondary to medications or other substances

Rare Disorders Cohort

Inclusion Criteria:

Participants who meet the following inclusion criteria are eligible for enrollment into this cohort:

1. Have an established Rare Coagulation Disorder (RCD) diagnosis of one of the following:

1. PAI-1 deficiency
2. Factor I, II, V, VII, X, XI, XIII deficiencies
3. Combined FV and FVIII deficiency
4. Plasminogen deficiency
5. Decreased tissue plasminogen activator
6. Afibrinogenemia/hypofibrinogenemia/dysfibrinogenemia
7. Thrombotic Thrombocytopenia Purpura or Congenital Hemolytic Uremic Syndrome
8. Wiskott-Aldrich
9. Methylenetetrahydrofolate Reductase Deficiency

Exclusion Criteria:

None

Bleeding NOS Cohort

Inclusion Criteria:

Participants who meet the following inclusion criteria are eligible for enrollment into this cohort:

1. Have a bleeding phenotype as indicated by an ISTH Bleeding Assessment Tool score of ≥4 for adult males, ≥6 for adult females, or ≥3 for children younger than 18 years with an unknown diagnosis, OR
2. Connective tissue disorder with bleeding tendency as indicated by an ISTH Bleeding Assessment Tool score of ≥4 for adult males, ≥6 for adult females, or ≥3 for children younger than 18 years.

Exclusion Criteria:

None

Thrombosis/Thrombophilia Cohort

Inclusion Criteria

Participants who meet the following inclusion criteria are eligible for enrollment into this cohort:

1. Have a prior history of arterial or venous thrombosis. 2. Participants with a known congenital or acquired thrombophilia with or without thrombosis.

a. Common congenital thrombophilias: i. Protein C deficiency ii. Protein S deficiency iii. Antithrombin deficiency iv. Factor V Leiden v. Prothrombin gene mutation b. Rare genetic factors i. Hyperhomocysteinemia c. Indeterminate genetic factors i. Elevated factor VIII ii. Elevated factor IX iii. Elevated factor XI iv. Elevated lipoprotein (a) d. Acquired thrombophilias i. Lupus anticoagulant ii. Anti-cardiolipin antibodies/Beta2 glycoprotein antibodies iii. Antiphospholipid syndrome

Exclusion Criteria Acquired thrombophilia secondary to medications (birth control pills or hormone replacement therapy), overweight or obesity, smoking, cancer, pregnancy, surgery, injury, prolonged inactivity/bedrest, heart failure, inflammatory bowel disease, or kidney disease

Non-Neoplastic Hematologic Conditions Cohort

Inclusion Criteria

Participants who meet the following inclusion criteria are eligible for enrollment into this cohort:

1. Having any congenital or acquired non-neoplastic hematologic disorder not included in any other cohort

Exclusion Criteria None

Arm/Module Participant Selection

Previously Untreated Patients Arm

Inclusion Criteria:

1. Diagnosis of congenital hemophilia A (FVIII <40%) or hemophilia B (FIX <40% or below lower limit for age)
2. Age <18 years at time of enrollment
3. Parent or authorized guardian or legally authorized representative (LAR) can provide informed consent
4. Care established at one of the ATHN Transcends participating HTCs
5. Clotting Factor Concentrate (CFC) exposure, fresh frozen plasma (FFP), cryoprecipitate, and single donor platelets <3 exposure days (ED)

Exclusion Criteria

1. Concomitant diagnosis with another bleeding disorder
2. History of a confirmed, positive inhibitor

INHIBIT Module

Inclusion Criteria:

1. Diagnosis of severe factor VIII deficiency with baseline factor VIII level <1% 2. Initiating or plan to initiate prophylaxis with emicizumab or factor replacement 3. Factor concentrate exposure, Fresh Frozen Plasma (FFP), cryoprecipitate, and single donor platelets ≤3 EDs 4. ≤5 years of age

Exclusion Criteria

1. Concomitant diagnosis with bleeding disorder other than hemophilia A
2. Immune disorder
3. Previous history or presence of factor VIII inhibitor. A confirmed, positive inhibitor is defined as two consecutive positive inhibitor titers (≥ 0.6 BU) that result in changes in treatment recommendations.

Efanesoctocog alfa (ALTUVIIIO®) Module

Inclusion criteria:

1. Ability of the potential participant's legally authorized representative (e.g., their parent or legal guardian) to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local participant privacy regulation.
2. People with severe HA with a baseline FVIII activity of less than 1%. (While inclusion for participation in ATHN Transcends lists <5% FVIII activity, this proposed module will limit enrollment to people with FVIII activity levels of <1%.) Other severities may be included per ATHN Transcends PI approval.
3. <18 years of age.
4. No history of a confirmed, positive FVIII inhibitor.
5. Sex assigned at birth of male, female, or intersex.
6. Participants should have no more than three (3) exposure days of blood products (fresh frozen plasma, cryoprecipitate, or platelets), no more than three (3) doses of any FVIII concentrate other than efanesoctocog alfa, and up to three (3) doses of efanesoctocog alfa prior to enrollment.
7. Site PI confirmed all inclusion criteria has been met.

Exclusion criteria:

1. Not meeting all the inclusion criteria; confirmed by site PI.
2. Any exposure to blood products or FVIII replacement products except as described in the inclusion criteria.
3. History of positive inhibitor testing.
4. History of hypersensitivity reactions associated with efanesoctocog alfa administration.
5. Other coagulation disorder(s) in addition to Hemophilia A.
6. Any concurrent clinically significant major disease such as cancer that, in the opinion of the investigator, would make the participant unsuitable for enrollment.
7. Concurrent systemic treatment with chemotherapy and/or other immunosuppressant medications. Use of corticosteroids for the treatment of asthma or management of acute allergic or otherwise life-threatening episodes is allowed except for systemic corticosteroid treatment given to children daily or on an alternate day schedule at > 2 mg/kg/day of prednisone or its equivalent or > 20 mg/day if the duration is longer than 14 days.
8. Enrollment in a concurrent clinical interventional drug study.
9. Intake of an Investigational Medicinal Product within three (3) months prior to inclusion in this study.
10. Inability to comply with study requirements.
11. Other, unspecified reasons that, in the investigator's opinion, make the participant unsuitable for enrollment.

Hemophilia Natural History Arm

Inclusion Criteria

1. Congenital or acquired hemophilia A or B of any severity with or without inhibitors receiving a current therapy, a non-factor product, or for whom use of a non-factor product is a possibility, OR
2. Females of any age, with confirmed congenital hemophilia A or B carrier status with genetic mutational analysis and any factor level.

Exclusion Criteria

1. Presence of any known bleeding disorder other than congenital hemophilia A or B
2. Presence of concurrent hemophilia and a second hemostatic defect (low von Willebrand Factor (vWF) without vWD diagnosis is not excluded)
3. Unable or unwilling to comply with the study arm protocol.

Nonacog beta pegol (Rebinyn®) Module

Inclusion Criteria:

1. Has provided signed written consent for the nonacog beta pegol (Rebinyn®)Module before any study-related activities.
2. Male participants, at any age with hemophilia B, naïve or minimally exposed (up to 3 EDs) to nonacog beta pegol treatment at time of study enrollment. Additional doses may be allowable per ATHN Transcends PI approval.
3. Decision to initiate continuous prophylaxis treatment with commercially available nonacog beta pegol has been made by the participant(s)/Legally Authorized Representative(s) (LAR(s)) and the treating physician before and independently from the decision to include the participant in this study.

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as having given informed consent in this study.
2. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation, including a diagnosis or suspicion of attention deficit hyperactivity disorder (ADHD) or autism spectrum disorder (ASD) per the discretion of the Principal Investigator.
3. Known or suspected hypersensitivity to nonacog beta pegol or related products.
4. Clinical suspicion or presence of FIX inhibitor at time of inclusion.
5. Inability or unwillingness to undergo neurological assessment/structured developmental history.

Emicizumab (Hemlibra®) Module

Inclusion Criteria:

1. Participant currently treated with emicizumab (Hemlibra®)
2. Currently enrolled in the Hemophilia Natural History Arm of ATHN Transcends

Exclusion Criteria:

1. Unable or unwilling to comply with the protocol

Distress Module

Inclusion Criteria:

1. Congenital hemophilia A or B of any severity with or without inhibitors receiving a current therapy, a non-factor product, or for whom use of a non-factor product is a possibility
2. Age 18 years of age or older
3. English speaking

Exclusion Criteria:

1. Presence of any known bleeding disorder other than congenital hemophilia A or B;
2. Presence of concurrent hemophilia and a second hemostatic defect (low von Willebrand Factor (vWF) without vWD diagnosis is not excluded); and
3. Unable or unwilling to comply with the study arm protocol

Hemophilia Gene Therapy Outcomes Arm

Inclusion Criteria

1. Hemophilia A or B of any severity with or without inhibitors having received or will receive a hemophilia gene transfer product in the next 6 months.
2. Age 18 years and older.
3. Able to give informed consent.

Exclusion Criteria None

Etranacogene dezaparvovec (HEMGENIX®) Module

Inclusion Criteria:

Etranacogene dezaparvovec (HEMGENIX®) Cohort

1. Age 18 years of age or older
2. Treatment with commercial etranacogene dezaparvovec (HEMGENIX®)
3. Have provided signed written informed consent within 3 months before or within 6 months after etranacogene dezaparvovec (HEMGENIX®) treatment, or within 6 months of when the study is initiated at the treating site.

FIX Prophylaxis Cohort

1. Age 18 years of age or older
2. Treatment with FIX prophylaxis therapy
3. Has provided signed written consent at any time for ATHN Transcends Study

Exclusion Criteria, both cohorts:

1. Have been treated with etranacogene dezaparvovec in a clinical trial prior to commercial availability. These patients are still eligible for enrollment in the Gene Therapy Outcomes Arm, and their data may be collected for separate analysis.

Congenital Platelet Disorders Arm

Inclusion Criteria

1. Platelet adhesion defect

   1. Bernard Soulier syndrome (Defective GPIb-IX-V receptor, impaired adhesion to vWF)
   2. Velocardio-facial syndrome/DiGeorge syndrome (Defective GPIb-IX-V receptor)
   3. Platelet type vWD (Defective GPIb-IX-V, gain of function interaction between vWF-GP1bα)
2. Platelet aggregation defect

   1. Glanzmann thrombasthenia (Defective integrin αIIbβ3 (GPIIb/IIIa)
   2. Platelet aggregation defect, NOS
3. Agonist receptor defects

   1. Epinephrine
   2. ADP
   3. Collagen
   4. Thromboxane A2
4. Platelet signaling defects

   1. Cyclooxygenase deficiency (PTGS1 mutation)
   2. Phospholipase A2 deficiency
   3. Thromboxane synthase deficiency (TBXAS1 mutation)
   4. G protein activation defect (GNAS mutation)
   5. Scott syndrome (defect in phosphatidyl serine translocation)
5. Platelet Granule disorders

   1. Dense granule storage pool disorder

      * Hermansky Pudlak syndrome
      * Chediak Higashi syndrome
      * Griscelli syndrome
   2. Alpha granule storage pool disorder

      * Grey platelet syndrome
      * Arthrogryposis-Renal Dysfunction-Cholestasis (ARC) syndrome
      * Quebec platelet disorder
      * Paris-Trousseau syndrome
   3. Combined alpha delta granule deficiency
6. Platelet cytoskeletal structure defects

   1. Wiskott Aldrich syndrome
   2. MYH9 associated disorders (myosin heavy chain)

      * May Hegglin syndrome
      * Fechtner syndrome
      * Sebastian syndrome
      * Epstein syndrome
   3. Other mutations

      * FLNA mutations (Filamin)
      * DIAPH1 (Actin and microtubules)
      * ACTN1 (alpha actinin)
      * TPM4 (tropomyosin)
      * TUBB1 (beta tubulin)
7. Other Congenital thrombocytopenias

   1. Familial platelet disorders and predisposition to AML (RUNX1)
   2. X linked thrombocytopenia with dyserythropoiesis (GATA1)
   3. Congenital amegakaryocytic thrombocytopenia (MPL)

Exclusion Criteria

1. Diagnosis of von Willebrand Disease (Meeting the definition of vWD or low vWF per most recent international guidelines)
2. Diagnosis of Hemophilia A or Hemophilia B (Factor VIII or IX ≤ 40%)

Glanzmann Thrombasthenia (GT) Module

Inclusion Criteria

1. Participant has signed the informed consent/assent form
2. Participant has flow cytometry or aggregometry or genetics confirmed GT
3. Participant is willing to perform study procedures, including daily bleed tracking for 3 months and further if requested
4. Participants are 2 years or older at time of consent

Exclusion Criteria None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a real-world study in which participants with congenital or acquired blood disorders will be enrolled.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2035-06 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
To determine the safety of therapies used in the treatment of participants with congenital or acquired non-neoplastic, bleeding and clotting disorders and connective tissue disorders with bleeding tendency (blood disorders). | 15 years
  Safety will be measured by those events in the European Safety Surveillance (EUHASS)1:
  1. Allergic or other acute events
  2. Treatment-emergent side effects of therapy
  3. Transfusion transmitted infections
  4. Inhibitor development
  5. Thrombosis
  6. Cardiovascular events
  7. Malignancies
  8. Neurological events
  9. Death
  In addition to the modified EUHASS endpoints, the following events will be collected as adverse events of special interest (AESI):
  1. The occurrence of thrombotic microangiopathies, injection site reactions and cases of potential drug-induced liver injury
  2. The development of anti-drug antibodies, to be measured and confirmed, if feasible
  3. Severe, unanticipated bleeding
  4. Hospitalizations
  5. Glomerulonephritis
  6. Any arm or module-specific AESI as stated in their corresponding Safety Assessment section
  Additional safety events of interest may be collected.

SECONDARY OUTCOMES:
To establish a platform to support study arms and modules for participants with blood disorders. | 15 years
  For each Arm, a brief set of data elements of interests will be developed and reported for study participants.
To describe medication dosing regimens in participants with blood disorders. | 15 years
  This objective will be evaluated by:
  1. Determining the number of participants who initiate and/or switch treatment with non-factor products and participants' reasons for initiating and/or switching treatment with non-factor products
  2. Determining the number of participants who do not initiate treatment with non-factor products
  3. Determining the number of participants who switch between different non-factor products and the participants' reasons for switching non-factor products
  4. Determining the number of participants who discontinue treatment with non-factor products and participants' reasons for discontinuing treatment with non-factor products
To describe real-world effectiveness of therapies used for participants with blood disorders. | 15 years
  1. Health care utilization as measured by number and type of visits and hospitalizations per year
  2. Patient reported outcomes (PROs) as measured by the Patient Reported Outcomes Measurement Information System (PROMIS®) Profile 29/25/Parent Proxy, Global Adherence Rating (GAR) (ages 7 and older), CATCH, and EQ-5D5L
To grow and evolve the ATHN Transcends Biorepository for current and future research through the collection of biospecimens from participants enrolled on this protocol | 15 years
  All participants have the option to provide consent to have specimens stored in the ATHN Transcends Biorepository. Samples will be collected as needed, including at the Baseline Visit, Annual Visit, and at Study Exit Visit (if not collected at your Annual Visit), as funding allows.
To describe bleeding events, changes in overall bleeding, and annualized bleeding rate (ABR) as measured by individual bleeding components. | 15 years
  This objective will be calculated per ISTH Bleeding Assessment Tool (ISTH BAT), participant completed Treatment and Bleed log, and if applicable, a Pictorial Bleeding Assessment Chart (PBAC), for relevant diagnoses.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Recht, MD, PhD, MBA, Principal Investigator — Yale University School of Medicine & National Bleeding Disorders Foundation; Tammuella Chrisentery-Singleton, MD, Principal Investigator — ATHN, Ochsner Clinic Foundation
Locations (71):
- United States (71):
  - Arizona Hemophilia and Thrombosis Treatment Center at Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Center for Bleeding Disorders, Little Rock, Arkansas
  - Orthopaedic Institute for Children HTC, Los Angeles, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University of California at Davis Hemophilia Treatment Center, Sacramento, California
  - Loma Linda Hemoglobinopathy and Inherited Bleeding Disorder Program, San Bernardino, California
  - Hemophilia & Thrombosis Treatment Center at UC San Diego Health, San Diego, California
  - Rady Children's Hospital San Diego, San Diego, California
  - University of California, San Francisco Hemophilia & Thrombosis Center, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale Hemophilia Treatment Center, New Haven, Connecticut
  - Delaware Hemophilia Treatment Center, Wilmington, Delaware
  - Georgetown University, Washington D.C., District of Columbia
  - Children's National Hemophilia Center, Washington D.C., District of Columbia
  - University of Florida Hemophilia Treatment Center, Gainesville, Florida
  - University of Miami Comprehensive Hemophilia Treatment Center, Miami, Florida
  - Arnold Palmer Hospital for Children - The Haley Center for Children's Cancer and Blood Disorders, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Hospital Center for Bleeding & Clotting Disorders, Tampa, Florida
  - Comprehensive Bleeding Disorders Center at Emory University and Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory/Children's Health Care of Atlanta, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - Iowa Hemophilia and Thrombosis Center, Iowa City, Iowa
  - Louisiana Center for Bleeding and Clotting Disorders, Tulane University, New Orleans, Louisiana
  - Maine Hemophilia and Thrombosis Center, Scarborough, Maine
  - Johns Hopkins University Hemophilia Treatment Center, Baltimore, Maryland
  - Massachusetts General Hospital Comprehensive Hemophilia and Thrombosis Treatment Center, Boston, Massachusetts
  - Central Michigan Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Health System Bleeding and Thrombosis Treatment Center, Detroit, Michigan
  - Mayo Comprehensive Hemophilia Center, Rochester, Minnesota
  - Children's Mercy Hospital - Kansas City, Kansas City, Missouri
  - The John Bouhasin Center for Children with Bleeding Disorders, St Louis, Missouri
  - Cure 4 The Kids Foundation, Las Vegas, Nevada
  - Hemostasis and Thrombosis Center of Nevada, Reno, Nevada
  - Newark Beth Israel Medical Center - Hemophilia Center, Newark, New Jersey
  - University of New Mexico Ted R. Montoya Hemophilia & Thrombosis Program, Albuquerque, New Mexico
  - Western New York BloodCare, Buffalo, New York
  - Northwell Health Hemostasis and Thrombosis Center at Long Island Jewish and Cohen Children's Medical Center, Hyde Park, New York
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - American Thrombosis and Hemostasis Network, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Comprehensive Hemophilia Treatment Center, University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - St. Jude Affiliate Clinic at Novant Health Hemby Children's Hospital, Charlotte, North Carolina
  - East Carolina University Hemophilia Treatment Center, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Akron Children's Hospital - Showers Center for Cancer & Blood Disorders, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Hemophilia & Thrombosis Center, Cincinnati, Ohio
  - University of Cincinnati Medical Center Hemophilia Treatment Center, Cincinnati, Ohio
  - University Hospitals Health System Cleveland, Cleveland, Ohio
  - Nationwide Children's Hospital Columbus, Columbus, Ohio
  - Dayton Children's Hemostasis and Thrombosis Center, Dayton, Ohio
  - Northwest Ohio Hemophilia Treatment Center at the Toledo Hospital, Toledo, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Penn Comprehensive Hemophilia and Thrombophilia Program/Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Hemostasis and Thrombosis Center, Providence, Rhode Island
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Children's Blood and Cancer Center of Central Texas, Austin, Texas
  - North Texas Hemophilia and Thrombosis Program - Pediatric Program / Center for Cancer & Blood Disorders, Dallas, Texas
  - North Texas Comprehensive Hemophilia Treatment Center, Dallas, Texas
  - Gulf States Hemophilia and Thrombophilia Center, Houston, Texas
  - Texas Children's Hemophilia & Thrombosis Center/Baylor College of Medicine, Houston, Texas
  - South Texas Comprehensive Hemophilia and Thrombophilia Treatment Center, San Antonio, Texas
  - Washington Center for Bleeding Disorders, Seattle, Washington
  - Hemophilia Outreach Center Green Bay, Green Bay, Wisconsin
  - Comprehensive Center for Bleeding Disorders, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weijer C, Freedman B, Fuks A, Robbins J, Shapiro S, Skrutkowska M. What difference does it make to be treated in a clinical trial? A pilot study. Clin Invest Med. 1996 Jun;19(3):179-83. PMID 8724821
- [Background] Braunholtz DA, Edwards SJ, Lilford RJ. Are randomized clinical trials good for us (in the short term)? Evidence for a "trial effect". J Clin Epidemiol. 2001 Mar;54(3):217-24. doi: 10.1016/s0895-4356(00)00305-x. PMID 11223318
- [Background] West J, Wright J, Tuffnell D, Jankowicz D, West R. Do clinical trials improve quality of care? A comparison of clinical processes and outcomes in patients in a clinical trial and similar patients outside a trial where both groups are managed according to a strict protocol. Qual Saf Health Care. 2005 Jun;14(3):175-8. doi: 10.1136/qshc.2004.011478. PMID 15933313
- [Background] Unger JM, Barlow WE, Martin DP, Ramsey SD, Leblanc M, Etzioni R, Hershman DL. Comparison of survival outcomes among cancer patients treated in and out of clinical trials. J Natl Cancer Inst. 2014 Mar;106(3):dju002. doi: 10.1093/jnci/dju002. Epub 2014 Mar 13. PMID 24627276
- [Background] https://www.fda.gov/drugs/resources-information-approved-drugs/hematologyoncology-cancer-approvals-safety-notifications. Accessed 04 Jul 2019
- [Background] https://www.clinicaltrials.gov/ct2/results?cond=Hematologic+Diseases&term=&cntry=&state=&city=&dist=. Accessed 04 Jul 2019
- [Background] Konkle BA, Recht M; members of Working Group 2, the NHLBI State of the Science Workshop on factor VIII inhibitors: Generating a national blueprint for future research. The national blueprint for 21st century data and specimen collection and observational cohort studies: NHLBI State of the Science Workshop on factor VIII inhibitors. Haemophilia. 2019 Jul;25(4):590-594. doi: 10.1111/hae.13772. PMID 31329362
- [Background] Iorio A, Keepanasseril A, Foster G, Navarro-Ruan T, McEneny-King A, Edginton AN, Thabane L; WAPPS-Hemo co-investigator network. Development of a Web-Accessible Population Pharmacokinetic Service-Hemophilia (WAPPS-Hemo): Study Protocol. JMIR Res Protoc. 2016 Dec 15;5(4):e239. doi: 10.2196/resprot.6558. PMID 27977390